CLINICAL TRIAL: NCT02511262
Title: Clinical Trial Protocol for the Illumigene® Mycoplasma Direct Assay
Brief Title: Detection of Mycoplasma Pneumoniae
Status: Completed | Type: Observational
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-DHF-309-004.001
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Mycoplasma Pneumoniae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dual throat swabs.

GROUPS / COHORTS (1):
- Specimen Collection: Prospective patients with symptoms of upper respiratory infections which may be attributable to Mycoplasma pneumoniae, or from patients suspected of having Mycoplasma pneumoniae.
  Interventions: Device: illumigene® Mycoplasma Direct, illumipro-10

INTERVENTIONS:
Device: illumigene® Mycoplasma Direct, illumipro-10 — DNA amplification assay

SUMMARY:
The objective of this Clinical Trial is to define the methods to be used to document that illumigene® Mycoplasma Direct meets its intended use claims, using the illumipro instrument, with throat swab samples collected from symptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject has willingly given written informed consent.
* Specimens provided from subjects with symptoms of upper respiratory infections which may be attributable to Mycoplasma pneumoniae, or from patients suspected of having Mycoplasma pneumoniae.
* Dual throat swab collected per subject.

Exclusion Criteria:

* Subjects who are unwilling to sign the written informed consent.
* Multiple sets of specimens collected from the same subject.
* Subjects who are unwilling or unable to provide the required number of throat swabs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective patients with symptoms of upper respiratory infections which may be attributable to Mycoplasma pneumoniae, or from patients suspected of having Mycoplasma pneumoniae.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of Mycoplasma Pneumoniae to aid in the diagnosis of M. pneumoniae infections. | Up to 14 days
  Testing of each enrolled subject's samples will be performed within 14 days of collection.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sacred Heart Health System, Pensacola, Florida
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Cook Children's Healthcare System (CCHCS), Fort Worth, Texas